CLINICAL TRIAL: NCT05991479
Title: Effect of Pilates Exercises on Muscle Strength and Balance After Healed Lower Limb Burns
Brief Title: Pilates Exercises on Muscle Strength and Balance After Healed Lower Limb Burns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmeen Hamada Lotfy Mohamed, Assistant Lecturer at Department of Surgery and Burn - Faculty of Physical Therapy - Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 286206
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Lower Limb Burns
Keywords: Pilates exercises; Muscle strength; Balance; Lower limb burns
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Pilates exercises plus traditional physical therapy programme) (Experimental): Pilates exercises: The Pilates training protocol will take 60 min per session, including 10 min of warm up prior to initiating the Pilates technique, 40 min for Pilates exercises and 10 min for cool down. The number of repetitions will be 10 times. The patient will perform the following Pilates exercises: (Hundred exercises, spine stretch, single leg stretch , double leg stretch, criss cross, swimming, one leg kick, side kick, clam, one leg circle, shoulder bridge, hip twist, roll up and down and standing footwork).Pilates training (3 sessions/week) for 8 weeks.
  traditional physical therapy programme: consisting of a supervised and individualized exercise programme for three sessions per week for eight weeks which will include:
  1. Stretching exercises for calf and hamstring muscles.
  2. Strengthening exercises for hip, knee, ankle, and foot muscles.
  3. Deep friction massage for scar management:
  Interventions: Other: Pilates exercises; Other: Traditional physical therapy programme:
- (traditional physical therapy programme) (Experimental): All patients will receive a traditional physical therapy programme consisting of a supervised and individualized exercise programme for three sessions per week for eight weeks which will include:
  1. Stretching exercises for calf and hamstring muscles.
  2. Strengthening exercises for hip, knee, ankle, and foot muscles.
  3. Deep friction massage for scar management:
  Interventions: Other: Traditional physical therapy programme:

INTERVENTIONS:
Other: Pilates exercises — Pilates exercises:
  The subjects will receive Pilates training (3 sessions/week) for 8 weeks. The Pilates training protocol will take 60 min per session, including 10 min of warm up prior to initiating the Pilates technique, 40 min for Pilates exercises and 10 min for cool down. The number of repetitions will be 10 times. The patient will perform the following Pilates exercises: (Hundred exercises, spine stretch, single leg stretch , double leg stretch, criss cross, swimming, one leg kick, side kick, clam, one leg circle, shoulder bridge, hip twist, roll up and down and standing footwork).
  Arms: (Pilates exercises plus traditional physical therapy programme)
Other: Traditional physical therapy programme: — All patients will receive a traditional physical therapy programme consisting of 45 minutes per session of a supervised and individualized exercise programme for three sessions per week for eight weeks which will include:
  Stretching exercises for calf and hamstring muscles. Strengthening exercises for hip, knee, ankle, and foot muscles. Deep friction massage for scar management.

SUMMARY:
The study will be carried out on 76 patients suffering from lower limb burns with TBSA ranging from 30% to 40%. The patients will be subdivided into two groups of equal number.

Group (A): (The study group) who will receive Pilates exercise in addition to traditional physical therapy programme in the form of stretching and strengthening exercises and deep friction massage for scar management.

Group (B): (The control group) who will receive traditional physical therapy programme only.

DETAILED DESCRIPTION:
1. subjects: The patients will be subdivided into two groups of equal number.

   Group A: (The study group):

   This group will be composed of 38 patients with lower limb burns. Patients will receive Pilates exercise in addition to a traditional physical therapy programme in the form of stretching exercises, strengthening exercises and deep friction massage for scar management (3 sessions per week) for 8 weeks.

   1.2 Group B: (The control group): This group will be composed of 38 patients with lower limb burns. Patients will receive a traditional physical therapy programme in the form of stretching exercises, strengthening exercises and deep friction massage for scar management (3 sessions per week) for 8 weeks.
2. Equipment:

Therapeutic equipment:

Therapeutic equipment and tools in this study will include the following:

a)Pilates exercises: The subjects will receive Pilates training (3 sessions/week) for 8 weeks. The Pilates training protocol will take 60 min per session, including 10 min of warm up prior to initiating the Pilates technique, 40 min for Pilates exercises and 10 min for cool down. The number of repetitions will be 10 times.

The patient will perform the following Pilates exercises:

1. Hundred exercises:

   Patients will be asked to lie in supine position with arms at their sides and knees bent up in the air, then position their knees and hips in 90-degree angles. Then will be instructed to curl their head and shoulders off the floor. The arms then move up and down slowly, initiating the movement from the shoulder joint. The subjects will inhale for a count of five and exhale for a count of five and this step will be repeated until reach 100 counts.
2. Spine stretch:

   Each patient will be asked to sit in a long sitting position with her legs extended out in front of his with hip-distance apart, feet dorsiflexed. As he inhaled, his arms should be stretched out in front of her with palms down then, Exhale and reach her feet; keeping his arms parallel to the floor and contract the abdominal muscles, then inhale and return to his starting position. Repeat 10 times.
3. Single leg stretch:

   Patients will be asked to lie on their back and bring chin to chest, lifting head and neck off mat. Bend right knee into chest and place left hand on right knee and right hand on right ankle. Extend left leg off mat in Pilates stance while keeping lower back on mat. Change legs and hand position. Inhale for 1 set (right and left) and exhale for 1 set.
4. Double leg stretch:

   Each patient will be asked to lie on their back and bring chin to chest keeping chin to chest, bend both knees into chest and places hands around ankles. Extend legs off mat in Pilates stance and arms behind head. Open arms to sides and circle them around to ankles again as knees bend in. Inhale as arms and legs bend and exhale as they extend.
5. Criss cross:

   Patients will be asked to keep their chin to chest and hands behind head, bend knees so legs form 90° angle above the mat. Bend right knee into chest and extend left leg in Pilates stance. Twist left elbow towards right knee and look behind right elbow. Pass through center, with legs bent at 90° angle above the mat and both sides of back on mat and repeat to other side. Inhale when in center and exhale on twist.
6. Swimming:

   Patients will be asked to lie on their stomach with legs extended together in Pilates stance and arms extended in front of head shoulder width apart. Lift upper back, right arm, and left leg, keeping arm and leg straight. Alternate lifting arms and legs, always lifting the opposite arm and leg together, while keeping upper back lifted off mat. Inhale for 10 counts and exhale for 10 counts.
7. One leg kick:

   Patients will be asked to lie in the prone position, closing the back of the legs to the same leg hamstring and firming the buttock while increasing their abdominal strength.
8. Side kick:

   Each patient will be asked to lie on his left side, his shoulders, hips, and ankles on the same line extended and his both legs slightly slide forward so he can see her toes. Support his head on left arm as he inhaled, kick with his right leg to the level of the hip twice while dorsi-flexing his foot. Then breathe out and relax. Repeat it 10 times for each leg.
9. Clam:

   Patients will be asked to lie on the side. Resting the head on the arm or hand, then bend hips to approximately 45 and knees at 90. Make sure that one hip is lying above the other. Upper leg upwards while keeping the feet in contact with one another.
10. One leg circle:

    Patients will be asked to bring their thighs as perpendicular to the floor as possible. Circle the leg down toward the mat, then out to the right, and finally back to center.
11. Shoulder bridge:

    Each patient will be asked to lie in the crock line position then gently raise their lower back until he is resting on his shoulder. Then breathe in and hold the position. In this position lift one heel off the floor, then breathe out and lower it down. Repeat 10 times for each side.
12. Hip twist:

    Patients will be asked to sit on a mat and extend their legs in front. The body should be in the same position as a V-up. Rotate the hips to the right side of the body and circle legs to the right and down.
13. Roll up & roll down:

    Each patient will be asked to lie flat on the mat, breathe in, dorsi-flex his feet and raise his arms to 90 degrees, then try to raise his head and shoulders from the mat then breathe out and relax. Repeat 10 times.
14. Standing footwork:

Patient will be in standing position in "V stance" While keeping the Pilates "V", the patients will be instructed to rise up on their toes as far as possible while keeping the heels together. Then they lowered to the ground while keeping their spine neutral. Then the patient will be instructed to perform a plié (bending at the hips and knees). The patient will be instructed to breathe in deeply after beginning the movement and breathe out when performing the movement.

(b) Traditional physical therapy programme:

All patients will receive a traditional physical therapy programme consisting of 45 minutes per session of a supervised and individualized exercise programme for three sessions per week for eight weeks which will include:

1. Stretching exercises for calf and hamstring muscles by using the hold relax technique:

   - To achieve this, the limb will be placed at its limit of range and an isometric contraction will be sustained (for 5 to 10 seconds), followed by a voluntary relaxation of the tightened muscles. The limb will then be passively moved into the new range and sustained the stretch for 30 seconds for 3 repetitions at each time.
2. Strengthening exercises for hip, knee, ankle, and foot muscles:

   * One repetition maximum test (1RM): The patients will be tested to determine the amount of weight or load that will be used during the first week (of the 8 weeks program) as baseline loads.
   * To improve strength, free weights will be used for all exercises. During the first week, 50 to 60% of their individual 1RM will be set as the starting weight. Then, from the second week to the sixth, the weight will be increased to 70%-75% of their individual 1RM. The training amplitude will be then raised to 80%-85% of their individual 1RM that will be continued through weeks 7 and 8, holding 5 seconds at the end of the range. (Number of repetitions: 3 sets,10 repetitions in each).
3. Deep friction massage for scar management:

Deep circular movement by the balls of the thumb and sufficient drag will be applied to mobilize the tissue; tension and shear force will be used first followed by lifting and skin rolling when tissues become more pliable.

Measuring equipment:

a)Lafayette hand-held dynamometer (HHD): Hand-held dynamometer (HHD) is a convenient, reliable and valid instrument for muscle strength assessment.

in this study, Lafayette manual muscle testing (model 01163 USA) will be used for objectively quantifying the maximum isometric muscle strength of knee extensors and knee flexors.

knee extensors and flexors will be assessed while participants will be in a sitting position, hips and knees 90° flexed. The dynamometer will be positioned above the ankle joint, on the anterior aspect of the shank for assessing knee extensors, or on the posterior aspect of the shank for measuring knee flexors (b) Berg balance scale (BBS): Berg Balance Scale (BBS) is one of the most widely used tools for balance assessment. this scale has been shown to be a valid and reliable measure of balance.

The BBS consists of 14 items and has a maximum possible score of 56 points. It uses an ordinal scoring system in which each detail is rated, 0 being the lowest and 4 being the highest level of function.

(c) Arabic version of lower extremity functional scale (LEFS): The Arabic version of lower extremity functional scale will be used to assess lower limb functions. LEFS is an excellent patient-reported outcome measure that can be used in clinical practice and for research purposes to assess the level of activity limitation. The validity, reliability, and responsiveness of the LEFS have been established for musculoskeletal disorders. LEFS has 20 items each scored on 0-4 Likert scale and the overall score on the scale is produced by summing scores on all items. LEFS scores range from 0 to 80 with higher score indicating better functional ability.

ELIGIBILITY:
Inclusion Criteria:

The patients were chosen under the following criteria:

* Patients of both genders participated in this study.
* The patients' age ranged from 20-40 years old.
* Patients with lower limb second degree burn (partial thickness of thermal injury).
* Total burned surface area (TBSA) ranged from 30% to 40% measured by the rule of nine.
* Patients began the training programme after complete wound healing.

Exclusion Criteria:

* The current study excluded the following patients:
* Patients with an open wound at or near the treatment site.
* Patients with chemical or electrical burns.
* Patients with inhalation injury.
* Patients with any limitation in lower limb range of motion.
* Patients with musculoskeletal disorders or deformities that would impair performance during training and tests.
* Patients with visual or auditory disorders.
* Patients with neurological disorders.
* Patients with psychiatric illness, severe behavior or cognitive disorders.
* Uncooperative patients.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Lafayette hand-held dynamometer: | 8 weeks
  The maximum isometric force of knee flexors and extensors will be measured before and after treatment period using Lafayette HHD. The MIF will be measured through an accommodating isometric "make" test, where participants applied maximal force against the examiner while a steady position was maintained. Participants will perform three, 5 seconds contractions for each muscle group with a 30 second rest after each trial and 5 minutes rest between muscle groups. The average force of the three testing trials will be computed for each muscle. The examiner encourages participants to do their best effort during measurement. Knee extensors and flexors are assessed while participants are in a sitting position, hips and knees 90° flexed. The dynamometer is positioned above the ankle joint, on the anterior aspect of the shank for assessing knee extensors, or on the posterior aspect of the shank for measuring knee flexors.
Berg balance scale: | 8 weeks
  it consists of 14 items representing functional movements common in everyday life. Some items require that the patient maintain positions of increasing difficulty, from sitting to standing on one leg. Other items evaluate the ability to perform specific tasks, such as reaching forward, turning around and picking up an object from the floor. Scoring is based on the ability to meet certain time or distance requirements and to perform the items independently. Each task is scored on a 5-point scale from 0 to 4, giving a maximum score of 56, which indicates balance ability within the normal range.

SECONDARY OUTCOMES:
Arabic version of Lower extremity functional scale | 8 weeks
  it was translated to the classical Arabic language to enhance the use of the scale in all Arabic-speaking countries.
  Lower extremity functional scale (LEFS) is a patient-reported measure to examine the functional status in the presence of lower extremity musculoskeletal problems. The LEFS consists of 20 items, with scores ranging from 0 (extreme difficulty/unable to perform activity) to 4 (no difficulty). The total score can be obtained by summing the scores of the individual items. The maximum score of 80 indicates no functional limitations and the minimum score of 0 indicates extreme limitations.

CONTACTS AND LOCATIONS:
Overall Officials: yasmeen hamada, Principal Investigator — Cairo University
Locations (1):
- Faculty of physical therapy, Giza, Egypt